CLINICAL TRIAL: NCT07082335
Title: Clinical Characteristics and Prognosis of Simultaneous Versus Delayed Resection for Synchronous Colorectal Liver Metastasis: A Nationwide Multicenter Study Utilizing Propensity Score Matching Analysis
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zhang Feng-Min, MD, Shanghai 10th People's Hospital
Other Study IDs: 25K10
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer (CRC) often metastasizes to the liver, with synchronous metastases observed in 20% of cases. Surgical resection is the primary treatment, but the impact of simultaneous and staged resections on clinical outcomes remains unclear. This study employs propensity score matching (PSM) in a nationwide survey to compare clinical characteristics, complications, and survival, providing valuable insights for optimizing the management of colorectal liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1) a histologically confirmed diagnosis of colorectal cancer with liver metastases; and 2) age ≥ 18 years

Exclusion Criteria:

1) extrahepatic metastases; and 2) ineligibility for curative surgical resection based on preoperative assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This nationwide multicenter retrospective cohort study enrolled colorectal cancer patients with simultaneous liver metastases treated at 18 tertiary hospitals in China between January 2019 and December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
overall survival | 2 years
postoperative complications | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People Hospital, Yanchang Road, Jingan District, Shanghai,, Shanghai, Jingan, China

IPD SHARING:
Plan to Share IPD: Undecided